CLINICAL TRIAL: NCT01293929
Title: Association of Circulating Chemerin Levels and Arterial Stiffness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korea University (Other)
Responsible Party: Hye Jin Yoo, Korea university
Other Study IDs: A102065-1011-1070100
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-01

CONDITIONS: Obesity; Atherosclerosis
MeSH Terms: conditions — Obesity; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Non- obese group
- Obese group

SUMMARY:
Chemerin is a novel adipokine that might provide a link between chronic inflammation and obesity. Pulse wave velocity(PWV) is a useful method for examining arterial stiffness, meaning early-stage atherosclerosis. Therefore, in the present study, the investigators examined the relationship between circulating chemerin and arterial stiffness measured using PWV in obese persons.

ELIGIBILITY:
Inclusion Criteria:

* Self referred persons for visiting routine medical check in our clinic

Exclusion Criteria:

* Malignancy
* Severe renal or hepatic disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obese and age, gender matched non-obese group who underwent a medical health check in the Korea University Guro hospital
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
The difference of serum chemerin level between obese and non-obese groups | at the time of initial enrollment (4weeks)
  serum chemerin levels of all participants were by determined by an enzyme-linked immunosorbent assay (ELISA) kit (Biovender Laboratory Medicine Inc., Modrice, Czech Republic)

SECONDARY OUTCOMES:
The correlation of serum chemerin levels with arterial stiffness | at the time of enrollment (4 weeks)
  Arterial stiffness was measure using a Colin Waveform Analyser (model BP-203RPE II; Colin, Komaki, Japan). It was expressed as branchial ankle pulswe wave velocity (baPWV)

CONTACTS AND LOCATIONS:
Locations (1):
- Hye Jin Yoo, Seoul, South Korea